CLINICAL TRIAL: NCT06005857
Title: Use of Paper- Versus Digital Application-based Exercises to Support the Rehabilitation of People Operated by a Palmar Plate for an Intra-articular Distal Radius Fracture. A Multidisciplinary, Prospective, Randomized, Single-blind, Controlled Trial
Brief Title: Paper- vs Digital Application-based Exercises to Support Rehabilitation After Osteosynthesis of Distal Radius Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Fribourgeois (Other)
Responsible Party: Principal Investigator, Estoppey Daniel, Principal Investigator, Hôpital Fribourgeois
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PhysiAppHFR
Record Dates: First submitted 2023-08-09; First posted 2023-08-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Distal Radius Fracture
Keywords: distal radius fracture; smartphone application; post-operative rehabilitation; open reduction and internal fixation; range of motion
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The group will receive standard hand therapy program + rehabilitation program sustained by the use of a digital application.
  Interventions: Other: Standard hand therapy + home digital application-based exercises
- Control group (Active Comparator): The control group will receive a standard hand therapy program + paper-based (standard) rehabilitation program.
  Interventions: Other: standard hand therapy + home paper-based exercises

INTERVENTIONS:
Other: Standard hand therapy + home digital application-based exercises — Standard post-operative hand rehabilitation and home digital application-based exercises
  Arms: Experimental group
Other: standard hand therapy + home paper-based exercises — Standard post-operative hand rehabilitation and home paper-based exercises
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the difference between the use of paper- versus application-based (smartphone application) exercises in the rehabilitation of intra-articular fractures of the distal radius at the Cantonal Hospital of Fribourg, Switzerland.

The operation itself will proceed as usual. However, the rehabilitation will be aided by exercises based either on a paper support or on a digital application (smartphone application), in addition to follow-up by a hand therapist.

The aim is to determine which support provides the best improvement in wrist mobility and function, and to speed up the return to work.

DETAILED DESCRIPTION:
The aims of this study are:

1. To measure range of motion (flexion and extension) of the wrist in usual post-operative hand therapy sustained by the use of a digital application-based home exercise program compared with usual post-operative hand therapy sustained by the use of paper-based (standard) home exercice program.
2. To measure the following variables in usual post-operative hand therapy sustained by the use of a digital application-based home exercise program compared with usual post-operative hand therapy sustained by the use of paper-based (standard) home exercice program:

   * Patient-Rated Wrist Evaluation score
   * Return to work
   * Retorn to leisure
   * Range of motion in pronation and supination, in radial deviation and ulnar deviation
   * Distal radio-ulnar joint stability
   * Grip strength
   * Key pinch strength
   * Tripod pinch strength
   * Fracture healing
   * Fracture displacement
   * Patient satisfaction with exercise support
   * Patient participation in rehabilitation

Co-primary endpoint: range of motion (ROM) of the wrist, i.e. measured in degrees in flexion and extension.

Secondary endpoints:

* Clinical scores Patient-Rated Wrist Evaluation (PRWE). The Patient-Rated Wrist Evaluation (PRWE) score is to be completed by the patient himself, validated in French and in German. Pain score is measured by 5 items and function is measured by 10 items. The total score is based on 100 points. The best score is 0 and the worst score is 100.
* Partial sick-leave stoppage
* Total sick-leave stoppage
* Return to principal leisure
* Range of motion in pronation and supination, in radial deviation and ulnar deviation
* Distal radio-ulnar joint stability (compared with the healthy side)
* Grip strength (Hydraulic hand dynamometer JAMAR®), i.e. measured in kilograms
* Key pinch strength (B&L Engineering® Pinch Gauge), i.e. measured in kilograms
* Tripod pinch strength (B&L Engineering® Pinch Gauge), i.e. measured in kilograms
* Fracture healing
* Fracture displacement
* Patient satisfaction with exercise support
* Patient participation in rehabilitation

This research is a national, interdisciplinary, prospective, single-blind (investigator), parallel-group (experimental study, level of evidence I), monocentric (conducted at the HFR Fribourg - Hôpital cantonal) study.

All patients will undergo the same operative procedure. Upon arrival to the operating room, patients will be placed in supine position, the injured limb resting on a hand table. Standard anesthetic axillary nerve will be applied. All the operation will do by an experienced hand surgeon having minimum 5 years of post-specialization clinical experience. A standard modified Henry approach will be done. The DRF will be reduced and fixed with a palmar plate (Aptus Adaptive II, Medartis®). The stability of the distal radio ulnar joint (DRUJ) will be tested after the radius fixation. If the DRUJ will be instable, the ulnar styloid fracture will be fixed (osteo suture (PDS wire) or screw fixation (Aptus CCS 1.7/2.2, Medartis®).

The study participants will be allocated (randomization) to either Group 1 (standard hand therapy + home smartphone application-based exercises) or Group 2 (standard hand therapy + home paper-based exercises). The two groups will be matched as good as possible in terms of total numbers of participants per group, age (18-40 years or 41-65 years) and type of work (non-manual work or manual work) in order to minimize any possible bias due to structural differences in both groups.

All patients will undergo the same postoperative splint immobilization (removable palmar custom splint) for 6 weeks.

Patients will be randomly assigned to receive either a standard hand therapy program + smartphone application-based exercises or a standard hand therapy program + paper-based exercises. The follow-up will consist of a one-to-one therapy session per week durung 12 for monitoring, i.e. range of motion, swelling, scar, eventual adverse event, and the way of practicing exercises. In-person sessions will be supervised by a therapist involved in the study, who is certified in hand rehabilitation. Moreover, each patient is expected to practice by himself a daily home exercises program consisting of mobilization of the (i) thumb and (ii) long fingers in flexion-extension and mobilization of the (iii) wrist in flexion-extension, radio-ulnar inclination and pro-supination. Each exercise will be performed in 3 sets of 15 repetitions, 5 times a day. Strengthening exercises (iv) will be added from the sixth week post-surgery. Each training session will last around 15 minutes, and be repeated after a three-hours break. They are standard exercises used in the treatment of DRF and validated by several guidelines. If necessary, the treatment will be pursued after 12 weeks.

Each patient will be asked to fill in a paper daily diary on the number of exercises performed (number of repetitions actually performed per set requested, how many times per day). They will also be asked to fill in the level of pain felt at that time. A satisfaction questionnaire will be completed at the end of the treatment concerning the support (digital vs paper) used.

At 6 and 12 weeks, the blinded surgeon (not aware of the therapy the patient is undergoing) will research any clinical or radiological adverse events.

At 6 and 12 weeks, a blinded independent observer (not aware of the therapy the patient is undergoing) will measure the values required to achieve the aims 1 and 2.

Aim 1 :

An independent observer who is not the surgeon will measure, at 6 and 12 weeks, range of motion (flexion and extension) of patients of both groups (Group 1, with standard hand therapy + home digital application-based exercises; Group 2, with standard hand therapy + home paper-based exercises) with photography (Figure 11) and with a goniometer.

Aim 2 :

Patients of both groups (Group 1, with standard hand therapy + home digital application-based exercises; Group 2, with standard hand therapy + home paper-based exercises), the following variables will be measured:

* Patient-Rated Wrist Evaluation (PRWE)
* Return to work
* Retorn to leisure
* Range of motion in pronation and supination, in radial deviation and ulnar deviation
* Distal radio-ulnar joint stability
* Grip strength
* Key pinch strength
* Tripod pinch strength
* Fracture healing
* Fracture displacement
* Patient satisfaction with exercise support
* Patient participation in rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* Complete intra-articular DRF (classification AO 23 C1, C2 or C3)
* Simple palmar operative approach
* Simple palmar plate fixation
* Age 18-65 years
* Worker
* Own either a smartphone or other wireless device
* Consent form signed
* French or German speaker

Exclusion Criteria:

* Extra-articular or partial-articular DRF
* Double/triple operative approaches needed
* Bilateral procedure
* Fracture aged than more of 2 weeks
* Patient refusal/no informed consent
* Inability to give informed consent
* Previous wrist injury or surgery
* Rheumatoid polyarthritis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Range of motion in flexion-extension | From enrollment to the end of treatment at 3 months
  Measurement (in degrees) of joint mobility using a goniometer

SECONDARY OUTCOMES:
Wrist fonction score | From enrollment to the end of treatment at 3 months
  Patient-Rated Wrist Evaluation score at 6 and 12 weeks after surgery.
  The Patient-Rated Wrist Evaluation score measure the pain score of all 5 items, measure the function score of all the 10 items. The total score the sum of pain and function scores. The best score is 0 and the worst score is 100.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas TM Mészaros, MD, Study Director — HFR Fribourg, Hôpital Cantonal
Locations (1):
- HFR Fribourg, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No
Data will be secured and anonymized, and analyzed only by the principal investigator.

REFERENCES:
- [Background] Lu C, Hu Y, Xie J, Fu Q, Leigh I, Governor S, Wang G. The Use of Mobile Health Applications to Improve Patient Experience: Cross-Sectional Study in Chinese Public Hospitals. JMIR Mhealth Uhealth. 2018 May 23;6(5):e126. doi: 10.2196/mhealth.9145. PMID 29792290
- [Background] Valdes K, Gendernalik E, Hauser J, Tipton M. Use of mobile applications in hand therapy. J Hand Ther. 2020 Apr-Jun;33(2):229-234. doi: 10.1016/j.jht.2019.10.003. Epub 2020 Apr 3. PMID 32253058
- [Background] Murfin M. Know your apps: an evidence-based approach to evaluation of mobile clinical applications. J Physician Assist Educ. 2013;24(3):38-40. doi: 10.1097/01367895-201324030-00008. PMID 24261171
- [Background] Wallace S, Clark M, White J. 'It's on my iPhone': attitudes to the use of mobile computing devices in medical education, a mixed-methods study. BMJ Open. 2012 Aug 24;2(4):e001099. doi: 10.1136/bmjopen-2012-001099. Print 2012. PMID 22923627
- [Background] Lyngcoln A, Taylor N, Pizzari T, Baskus K. The relationship between adherence to hand therapy and short-term outcome after distal radius fracture. J Hand Ther. 2005 Jan-Mar;18(1):2-8; quiz 9. doi: 10.1197/j.jht.2004.10.008. PMID 15674780
- [Background] Wakefield AE, McQueen MM. The role of physiotherapy and clinical predictors of outcome after fracture of the distal radius. J Bone Joint Surg Br. 2000 Sep;82(7):972-6. doi: 10.1302/0301-620x.82b7.10377. PMID 11041584
- [Background] Brehmer JL, Husband JB. Accelerated rehabilitation compared with a standard protocol after distal radial fractures treated with volar open reduction and internal fixation: a prospective, randomized, controlled study. J Bone Joint Surg Am. 2014 Oct 1;96(19):1621-30. doi: 10.2106/JBJS.M.00860. PMID 25274787
- [Background] Kay S, McMahon M, Stiller K. An advice and exercise program has some benefits over natural recovery after distal radius fracture: a randomised trial. Aust J Physiother. 2008;54(4):253-9. doi: 10.1016/s0004-9514(08)70004-7. PMID 19025505
- [Background] Christensen OM, Kunov A, Hansen FF, Christiansen TC, Krasheninnikoff M. Occupational therapy and Colles' fractures. Int Orthop. 2001;25(1):43-5. doi: 10.1007/s002640000183. PMID 11374267
- [Background] Ezzat A, Baliga S, Carnegie C, Johnstone A. Volar locking plate fixation for distal radius fractures: Does age affect outcome? J Orthop. 2016 Feb 22;13(2):76-80. doi: 10.1016/j.jor.2016.01.001. eCollection 2016 Jun. PMID 27053837
- [Background] Mattila VM, Huttunen TT, Sillanpaa P, Niemi S, Pihlajamaki H, Kannus P. Significant change in the surgical treatment of distal radius fractures: a nationwide study between 1998 and 2008 in Finland. J Trauma. 2011 Oct;71(4):939-42; discussion 942-3. doi: 10.1097/TA.0b013e3182231af9. PMID 21986738
- [Background] Al Khudairy A, Hirpara KM, Kelly IP, Quinlan JF. Conservative treatment of the distal radius fracture using thermoplastic splint: pilot study results. Eur J Orthop Surg Traumatol. 2013 Aug;23(6):647-50. doi: 10.1007/s00590-012-1042-8. Epub 2012 Jul 14. PMID 23412175
- [Background] Jerrhag D, Englund M, Karlsson MK, Rosengren BE. Epidemiology and time trends of distal forearm fractures in adults - a study of 11.2 million person-years in Sweden. BMC Musculoskelet Disord. 2017 Jun 2;18(1):240. doi: 10.1186/s12891-017-1596-z. PMID 28576135
- [Background] Court-Brown CM, Caesar B. Epidemiology of adult fractures: A review. Injury. 2006 Aug;37(8):691-7. doi: 10.1016/j.injury.2006.04.130. Epub 2006 Jun 30. PMID 16814787